| l | |
|---|---|
| 2 | |
| 3 | STUDY OF ADULT STRABISMUS |
| 4 | (SAS1) |
| 5 | |
| 6 | A Prospective Observational Study of Adult |
| 7 | Strabismus |
| 8 | |
| 9 | SAS1a: A Prospective Observational Study of Adult Convergence Insufficiency (CI) |
| 10 | SAS1b: A Prospective Observational Study of Adult Divergence Insufficiency (DI) |
| 11 | SAS1c: A Prospective Observational Study of Adult Small-Angle Hypertropia (HT) |
| 12 | |
| 13 | |
| 14 | PROTOCOL |
| 15 | |
| 16 | Version 2.0 |
| 17 | April 11, 2016 |
| 18 | |
| 19<br>20 | |
| 21 | |
| 22 | |
| 23 | |
| 24 | |
| 25 | |
| 26<br>27 | |
| 28 | |
| 29 | |
| 30 | |
| 31 | |
| 32 | |

# A PROSPECTIVE OBSERVATIONAL STUDY OF ADULT STRABISMUS (SAS1)

# 33 34 35

# PROTOCOL AMENDMENT I (4-11-16)

36 37

38

39

40

41

# **Proposed Change #1**

# **Current Protocol**

- Enrollment visit: Questionnaires and the symptom survey (if applicable) should be administered to the subject prior to other examination procedures.
- Follow-up visits: No specific mention regarding order of testing with respect to questionnaires and the symptom survey.

42 43 44

45

46

47

48

49

### **Proposed Change**

- Enrollment visit: Remove specific language regarding order of testing to allow questionnaires and the symptom survey (if applicable) to be completed at any time during the enrollment visit.
- Follow-up visits: Add specific language regarding order of testing at follow-up visits to require questionnaires and the symptom survey (if applicable) to be completed prior to testing.

50 51

52

53

54 55

# Rationale for Change

At the time of enrollment, treatment has not yet been initiated, therefore having knowledge of clinical assessments prior to completion of the questionnaires and the symptom survey is not expected to introduce any bias. In contrast, the questionnaires and symptom survey should be completed prior to clinical testing at any follow-up visit.

56 57 58

#### **Proposed Change #2**

- Current Protocol For subjects enrolled with Divergence Insufficiency
  - Distance esodeviation of 2 PD to 30 PD and at least 50% greater than at near by PACT

60 61 62

63

64

59

#### Proposed Change – For subjects enrolled with Divergence Insufficiency

- Distance esodeviation of 2 PD to 30 PD and distance deviation is at least 1.25 times (25% larger
- than) near deviation by PACT (i.e., maximum near deviation is at least 20% smaller than
- 65 distance deviation). The distance deviation must exceed the near deviation by at least the 66 amounts provided in the table below.

67 68

#### **PACT Values for DI Eligibility**

| Distance<br>Deviation | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 12 | 14 | 16 | 18 | 20 | 25 | 30 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| *Max Near<br>Deviation | 1 | 2 | 3 | 4 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 12 | 14 | 16 | 20 | 20 |

69 70 Calculation: Distance  $\geq$  Near x 1.25 or Near  $\leq$  Distance x 0.8

71 72

73

#### Rationale for Change

- The previous DI definition was developed by the SAS1 Planning Committee after literature 74 review and chart reviews. After the study started, the Strabismus Steering Committee has
- 75 lowered the threshold based on feedback from SAS1 investigators.

<sup>\*</sup>Near deviation is the nearest study-permitted prism based on Strabismus Procedures Manual.

76 77 78 **CONTACT INFORMATION** 79 80 81 **COORDINATING CENTER** 82 Raymond T. Kraker, M.S.P.H. (Director) 83 Jaeb Center for Health Research 84 15310 Amberly Drive, Suite 350 Tampa, FL 33647 85 Phone (888) 79PEDIG or (813) 975-8690 86 87 Fax (888) 69PEDIG or (813) 975-8761 88 Email: pedig@jaeb.org 89 90 PROTOCOL CHAIR 91 92 Eric Crouch, M.D. Virginia Pediatric Eye Center 93 94 880 Kempsville Road, Suite 2500 95 Norfolk, VA 23502 Phone (757) 461-0050 96 97 Fax (757) 461-4538 Email: ercrouch@virginiapediatriceye.com 98

# TABLE OF CONTENTS

| 102 | 100 | TABLE OF CONTENTS | |
|---|---|---|---|
| 103 | | CIVA DEED 4. DA CIVOD CANDA AND CAND | |
| 1.04 | | | |
| 105 | | | |
| 106 | | | |
| 107 | | | |
| 1.5.1 Synopsis of Study Design for CI | | • | |
| 109 | | | |
| 110 | | | |
| 111 1.5.4 Sludy Flow Chart: DL. 1 112 1.5.5 Synopsis of Study Design for HT 1 113 1.5.6 Study Flow Chart: HT. 1-1 114 CHAPTER 2: SUBJECT ENROLLMENT 2-1 115 2.1 Eligibility Assessment and Informed Consent 2-1 116 2.2 Eligibility Criteria for Cl. 2-1 117 2.2.1 Eligibility Criteria for DI 2-1 118 2.2.2 Eligibility Criteria for DI 2-1 119 2.2.3 Eligibility Criteria for HT 2-1 120 2.3 Historical Information 2-1 121 2.4 Procedures at the Enrollment Visit 2-1 122 2.4.1 Enrollment Procedures for CI 2-1 123 2.4.2 Enrollment Procedures for HT 2-1 124 2.4.3 Enrollment Procedures for HT 2-1 125 CHAPTER 3: TREATMENT AND FOLLOW-UP 3 126 3.1 Treatment 3 127 3.2 Visit Schedule 3 3.3 1 Flolow-up | | | |
| 112 1.5.5 Synopsis of Study Design for HT 1. 113 1.5.6 Study Flow Chart: HT 1-1 114 CHAPTER: SUBLECT EXBOLLMENT 2-1 115 2.1 Eligibility Assessment and Informed Consent 2-1 116 2.2 Eligibility Criteria for CI 2-1 117 2.2.1 Eligibility Criteria for DI 2-1 118 2.2.2 Eligibility Criteria for DI 2-1 119 2.2.3 Eligibility Criteria for DI 2-1 120 2.3 Historical Information 2-1 121 2.4 Procedures at the Enrollment Visit 2-1 122 2.4.1 Enrollment Procedures for CI 2-1 123 2.4.2 Enrollment Procedures for HT 2-1 124 2.4.3 Enrollment Procedures for HT 2-1 125 CHAPTER 3: TREATMENT AND FOLLOW-UP 3 126 3.1 Treatment 3 127 3.2 Visit Schedule 3 128 3.3 Follow-up Visit Testing Procedures for CI. 3 130 | | | |
| 113 1.5.6 Study Flow Chart: HT | | | |
| 114 CHAPTER 2: SUBJECT ENROLLMENT 2-1 115 2.1 Eligibility Assessment and Informed Consent 2-1 116 2.2 Eligibility Criteria (C.) 2-1 117 2.2.1 Eligibility Criteria for Cl 2-1 118 2.2.2 Eligibility Criteria for Dl 2-1 119 2.2.3 Eligibility Criteria for HT 2-1 120 2.3 Historical Information 2-1 121 2.4 Procedures at the Enrollment Visit. 2-1 122 2.4.1 Enrollment Procedures for Cl 2-1 123 2.4.2 Enrollment Procedures for Dl 2-1 124 2.4.3 Enrollment Procedures for Dl 2-1 125 CHAPTER 3: TREATMENT AND FOLLOW-UP 3-1 126 3.1 Treatment 3-1 127 3.2 Visit Schedule 3-3 128 3.3 Follow-up Visit Testing Procedures for Cl 3-3 129 3.3.1 Follow-up Visit Testing Procedures for Dl 3-3 130 3.3.2 Follow-up Visit Testing Procedures for Dl 3-3 131 3.3.3 Follow-up Visit Testing Procedures for HT 3-3 | | , 1 | |
| 115 2.1 Eligibility Assessment and Informed Consent 2-1 116 2.2 Eligibility Criteria for CI 2-1 118 2.2.1 Eligibility Criteria for DI 2-1 119 2.2.3 Eligibility Criteria for HT 2-1 120 2.3 Historical Information 2-1 121 2.4 Procedures at the Enrollment Visit 2-1 122 2.4.1 Enrollment Procedures for DI 2-1 123 2.4.2 Enrollment Procedures for DI 2-1 124 2.4.3 Enrollment Procedures for DI 2-1 125 CHAPTER 3: TREATMENT AND FOLLOW-UP 3 126 3.1 Treatment 3 127 3.2 Visit Schedule 3 128 3.3 Follow-up Visit Testing Procedures for CI 3 130 3.2.1 Follow-up Visit Testing Procedures for GI 3 131 3.3.1 Follow-up Visit Testing Procedures for H 3 132 3.4 Non-study Visit 3 <tr< td=""><td></td><td></td><td></td></tr<> | | | |
| 116 2.2 Eligibility and Exclusion Criteria 2-1 117 2.2.1 Eligibility Criteria for CI 2-1 118 2.2.2 Eligibility Criteria for DI 2-1 119 2.2.3 Eligibility Criteria for HT 2-1 120 2.3 Historical Information 2-1 121 2.4 Procedures at the Enrollment Visit. 2-1 122 2.4.1 Enrollment Procedures for CI 2-1 123 2.4.2 Enrollment Procedures for DI 2-1 124 2.4.3 Enrollment Procedures for DI 3-1 125 CHAPTER 3: TREATMENT AND FOLLOW-UP 3-3 126 3.1 Treatment 3-3 127 3.2 Visit Schedule 3-3 128 3.3 Follow-up Visit Testing Procedures for CI 3-3 129 3.3.1 Follow-up Visit Testing Procedures for CI 3-3 130 3.3.2 Follow-up Visit Testing Procedures for HT 3-3 131 3.3.3 Follow-up Visit Testing Procedures for HT 3-3 132 3.4 Non-study Visits < | | | |
| 117 2.2.1 Éligibility Criteria for CI 2-1 118 2.2.2 Eligibility Criteria for DI 2-1 119 2.2.3 Historical Information 2-1 120 2.3 Historical Information 2-1 121 2.4 Procedures at the Enrollment Visit. 2-1 122 2.4.1 Enrollment Procedures for CI 2-1 123 2.4.2 Enrollment Procedures for DI 2-1 124 2.4.3 Enrollment Procedures for HT 2-1 125 CHAPTER 3: TREATMENT AND FOLLOW-UP 3 126 3.1 Treatment 3 127 3.2 Visit Schedule 3 128 3.3 Follow-up Visit Testing Procedures (10-week and 12-month visits) 3 129 3.3.1 Follow-up Visit Testing Procedures for CI 3 130 3.2.2 Follow-up Visit Testing Procedures for DI 3 131 3.3.3 Follow-up Visit Testing Procedures for DI 3 132 3.4 Non-study Visits 3 133 3.5 Initiating a New Treatment 3 </td <td>_</td> <td>÷ .</td> <td></td> | _ | ÷ . | |
| 118 2.2.2 Eligibility Criteria for DI 2-1 119 2.2.3 Eligibility Criteria for HT 2-1 120 2.3 Historical Information 2-1 121 2.4 Procedures at the Enrollment Visit 2-1 122 2.4.1 Enrollment Procedures for CI 2-1 123 2.4.2 Enrollment Procedures for DI 2-1 124 2.4.3 Enrollment Procedures for HT 2-1 125 CHAPTER 3: TREATMENT AND FOLLOW-UP 3 126 3.1 Treatment 3 127 3.2 Visit Schedule 3 128 3.3 Follow-up Visit Testing Procedures (10-week and 12-month visits) 3 129 3.3.1 Follow-up Visit Testing Procedures for CI. 3 130 3.3.2 Follow-up Visit Testing Procedures for DI. 3 131 3.3.3 Follow-up Visit Testing Procedures for DI. 3 132 3.4 Non-study Visits 3 133 3.5 Initiating a New Treatment 3 132 4.1 Contacts by the Jack Center for Health Rese | | | |
| 119 2.2.3 Eligibility Criteria for HT 2-1 120 2.3 Historical Information 2-1 121 2.4 Procedures at the Enrollment Visit 2-1 122 2.4.1 Enrollment Procedures for Cl 2-1 123 2.4.2 Enrollment Procedures for Dl 2-1 124 2.4.3 Enrollment Procedures for HT 2-1 125 CHAPTER 3: TREATMENT AND FOLLOW-UP 3 126 3.1 Treatment 3 127 3.2 Visit Schedule 3 128 3.3 Follow-up Visit Testing Procedures (10-week and 12-month visits) 3 129 3.3.1 Follow-up Visit Testing Procedures for Cl 3 130 3.2.2 Follow-up Visit Testing Procedures for HT 3 131 3.3.3 Follow-up Visit Testing Procedures for HT 3 132 3.4 Non-study Visits 3 133 3.5 Initiating a New Treatment 3 134 CHAPTER 4: MISCELLANEOUS CONSIDERATIONS 4 135 4.1 Contacts by the Jaeb Center for Health Research and Sites 4 146 4.2 Subject Withdrawals 4 147 4.3 Management of Refractive Error 4 | | | |
| 120 2.3 Historical Information 2-1 2.4 Procedures at the Enrollment Visit. 2-1 2.4 Procedures at the Enrollment Visit. 2-1 2.4 Enrollment Procedures for CI 2-1 2.4 2.4.1 Enrollment Procedures for DI 2-1 2.4 2.4.3 Enrollment Procedures for DI 2-1 2.4.3 Enrollment Procedures for HT 2-1 2.4.3 Enrollment Procedures for HT 3.1 2-1 2.4.3 Enrollment Procedures for HT 3.1 3.2 CHAPTER 3: TREATMENT AND FOLLOW-UP 3.3 3.2 Visit Schedule 3.3 Follow-up Visit Testing Procedures (10-week and 12-month visits) 3.3 3.3 Follow-up Visit Testing Procedures for CI 3.3 3.3 Follow-up Visit Testing Procedures for DI 3.3 3.3 Follow-up Visit Testing Procedures for HT 3.3 3.3 Follow-up Visit Testing Procedures for HT 3.3 3.3 Follow-up Visit Testing Procedures for HT 3.3 3.5 Initiating a New Treatment 3.3 3.5 Initiating a New Treatment 3.3 3.5 Initiating a New Treatment 3.3 4.4 CHAPTER 4: MISCELLANEOUS CONSIDERATIONS 4.4 Contacts by the Jaeb Center for Health Research and Sites 4.2 Subject Withdrawals 4.4 4.5 Subject Withdrawals 4.4 Risks 4.5 Risk Assessment 4.5 Ris | _ | | |
| 121 2.4 Procedures at the Enrollment Visit. 2-1 122 2.4.1 Enrollment Procedures for CI. 2-1 123 2.4.2 Enrollment Procedures for DI. 2-1 124 2.4.3 Enrollment Procedures for HT. 2-1 125 CHAPTER 3: TREATMENT AND FOLLOW-UP. 3 126 3.1 Treatment. 3 127 3.2 Visit Schedule. 3 128 3.3 Follow-up Visit Testing Procedures (10-week and 12-month visits). 3 129 3.3.1 Follow-up Visit Testing Procedures for CI. 3 130 3.3.2 Follow-up Visit Testing Procedures for DI. 3 131 3.3.3 Follow-up Visit Testing Procedures for HT 3 132 3.4 Non-study Visits 3 133 3.5 Initiating a New Treatment 3 134 CHAPTER 4: MISCELLANEOUS CONSIDERATIONS. 4 4 4.1 Contacts by the Jaeb Center for Health Research and Sites 4 4.1 4.2 Subject Withdrawals 4 4.2 Subject Withdrawals 4 4.3 4.7 Risks 4.4 4.8 Kisks 4.4 4.5 Reporting of Adve | | | |
| 122 2.4.1 Enrollment Procedures for DI 2-1 123 2.4.2 Enrollment Procedures for DI 2-1 124 2.4.3 Enrollment Procedures for HT 2-1 125 CHAPTER 3: TREATMENT AND FOLLOW-UP 3 126 3.1 Treatment 3 127 3.2 Visit Schedule 3 128 3.3 Follow-up Visit Testing Procedures (10-week and 12-month visits) 3 129 3.3.1 Follow-up Visit Testing Procedures for CI 3 130 3.3.2 Follow-up Visit Testing Procedures for DI 3 131 3.3.3 Follow-up Visit Testing Procedures for HT 3 132 3.4 Non-study Visits 3 133 3.5 Initiating a New Treatment 3 134 CHAPTER 4: MISCELLANEOUS CONSIDERATIONS 4 135 4.1 Contacts by the Jaeb Center for Health Research and Sites 4 4 4.2 Subject Withdrawals 4 136 4.2 Subject Withdrawals 4 137 4.3 Management of Refractive Error 4 148 4.4 Risks of Examination Procedures 4 140 4.5 Reporting of Adverse Events 4 | _ | | |
| 123 2.4.2 Enrollment Procedures for DI 2-1 124 2.4.3 Enrollment Procedures for HT 2-1 125 CHAPTER 3: TREATMENT AND FOLLOW-UP 3 126 3.1 Treatment 3 127 3.2 Visit Schedule 3 128 3.3 Follow-up Visit Testing Procedures (10-week and 12-month visits) 3 129 3.3.1 Follow-up Visit Testing Procedures for CI 3 130 3.3.2 Follow-up Visit Testing Procedures for DI 3 131 3.3.3 Follow-up Visit Testing Procedures for HT 3 132 3.4 Non-study Visits 3 133 3.5 Initiating a New Treatment 3 134 CHAPTER 4: MISCELLANEOUS CONSIDERATIONS 4 135 4.1 Contacts by the Jaeb Center for Health Research and Sites 4 136 4.2 Subject Withdrawals 4 137 4.3 Management of Refractive Error 4 148 4.4 Risk Assessment 4 149 4.5 Reporting of Adverse Events 4 | | | |
| 124 2.4.3 Enrollment Procedures for HT. 2-1 125 CHAPTER 3: TREATMENT AND FOLLOW-UP. 3 126 3.1 Treatment. 3. 127 3.2 Visit Schedule. 3. 128 3.3 Follow-up Visit Testing Procedures (10-week and 12-month visits). 3. 129 3.3.1 Follow-up Visit Testing Procedures for CI. 3. 130 3.3.2 Follow-up Visit Testing Procedures for DI. 3. 131 3.3.3 Follow-up Visit Testing Procedures for HT. 3. 132 3.4 Non-study Visits. 3. 133 3.5 Initiating a New Treatment. 3. 134 CHAPTER 4: MISCELLANEOUS CONSIDERATIONS. 4. 135 4.1 Contacts by the Jaeb Center for Health Research and Sites. 4. 136 4.2 Subject Withdrawals. 4. 137 4.3 Management of Refractive Error. 4. 138 4.4 Risks. 4. 149 4.5.1 Risk Assessment. 4. 140 4.5 Reporting of Adverse Events. 4. 141 4.5.1 Risk Assessment. 4. 142 4.6 Discontinuation of Study. 4. 4.4 | | | |
| 125 CHAPTER 3: TREATMENT AND FOLLOW-UP 3 126 3.1 Treatment 3 127 3.2 Visit Schedule 3 128 3.3 Follow-up Visit Testing Procedures (10-week and 12-month visits) 3 129 3.3.1 Follow-up Visit Testing Procedures for CI 3 130 3.3.2 Follow-up Visit Testing Procedures for DI 3 131 3.3.3 Follow-up Visit Testing Procedures for HT 3 132 3.4 Non-study Visits 3 133 3.5 Initiating a New Treatment 3 134 CHAPTER 4: MISCELLANEOUS CONSIDERATIONS 4 4.1 Contacts by the Jaeb Center for Health Research and Sites 4 4.2 Subject Withdrawals 4 4.3 4.3 Management of Refractive Error 4 4.8 4.4 Risks 4 4.9 4.4.1 Risk Assessment 4 4.0 4.5.1 Risk Assessment 4 4.4.2 4.6 Discontinuation of | | | |
| 126 3.1 Treatment 3. 127 3.2 Visit Schedule 3. 128 3.3 Follow-up Visit Testing Procedures (10-week and 12-month visits) 3. 129 3.3.1 Follow-up Visit Testing Procedures for CI 3. 130 3.3.2 Follow-up Visit Testing Procedures for DI 3. 131 3.3.3 Follow-up Visit Testing Procedures for HT 3. 132 3.4 Non-study Visits 3. 133 3.5 Initiating a New Treatment 3. 134 CHAPTER 4: MISCELLANEOUS CONSIDERATIONS 4. 4 135 4.1 Contacts by the Jaeb Center for Health Research and Sites 4. 136 4.2 Subject Withdrawals 4. 137 4.3 Management of Refractive Error 4. 148 4.4 Risks 4. 138 4.4.1 Risks of Examination Procedures 4. 4.4.1 Risk Assessment 4. 140 4.5 Reporting of Adverse Events 4. 141 4.5.1 Risk Assessment 4. 14 | | 2.4.3 Enrollment Procedures for HT | 2-16 |
| 127 3.2 Visit Schedule 3. 128 3.3 Follow-up Visit Testing Procedures (10-week and 12-month visits) 3. 129 3.3.1 Follow-up Visit Testing Procedures for CI 3. 130 3.3.2 Follow-up Visit Testing Procedures for DI 3. 131 3.3.3 Follow-up Visit Testing Procedures for HT 3. 132 3.4 Non-study Visits 3. 133 3.5 Initiating a New Treatment 3. 134 CHAPTER 4: MISCELLANEOUS CONSIDERATIONS 4. 4.1 Contacts by the Jacb Center for Health Research and Sites 4. 4.2 Subject Withdrawals 4. 136 4.2 Subject Withdrawals 4. 137 4.3 Management of Refractive Error 4. 138 4.4 Risks 4. 139 4.4.1 Risk of Examination Procedures 4. 140 4.5 Reporting of Adverse Events 4. 141 4.5.1 Risk Assessment 4. 142 4.6 Discontinuation of Study 4. 143 <td></td> <td></td> <td></td> | | | |
| 128 3.3 Follow-up Visit Testing Procedures (10-week and 12-month visits) 3 129 3.3.1 Follow-up Visit Testing Procedures for CI 3 130 3.3.2 Follow-up Visit Testing Procedures for DI 3 131 3.3.3 Follow-up Visit Testing Procedures for HT 3 132 3.4 Non-study Visits 3 133 3.5 Initiating a New Treatment 3 134 CHAPTER 4: MISCELLANEOUS CONSIDERATIONS 4 135 4.1 Contacts by the Jaeb Center for Health Research and Sites 4 136 4.2 Subject Withdrawals 4 137 4.3 Management of Refractive Error 4 138 4.4 Risks 4 139 4.4.1 Risks of Examination Procedures 4 140 4.5 Reporting of Adverse Events 4 141 4.5.1 Risk Assessment 4 142 4.6 Discontinuation of Study 4 143 4.7 Travel Reimbursement 4 144 4.8 Study Costs 4 <t< td=""><td>-</td><td></td><td></td></t<> | - | | |
| 129 3.3.1 Follow-up Visit Testing Procedures for CI 3. 130 3.3.2 Follow-up Visit Testing Procedures for DI 3. 131 3.3.3 Follow-up Visit Testing Procedures for HT 3. 132 3.4 Non-study Visits 3. 133 3.5 Initiating a New Treatment 3. 134 CHAPTER 4: MISCELLANEOUS CONSIDERATIONS 4. 135 4.1 Contacts by the Jaeb Center for Health Research and Sites 4. 136 4.2 Subject Withdrawals 4. 137 4.3 Management of Refractive Error 4. 138 4.4 Risks 4. 139 4.4.1 Risks of Examination Procedures 4. 140 4.5 Reporting of Adverse Events 4. 141 4.5.1 Risk Assessment 4. 142 4.6 Discontinuation of Study 4. 143 4.7 Travel Reimbursement 4. 144 4.8 Study Costs 4. 145 4.9 General Considerations 4. 147 | | | |
| 130 3.3.2 Follow-up Visit Testing Procedures for DI | | | |
| 131 3.3.3 Follow-up Visit Testing Procedures for HT 3. 132 3.4 Non-study Visits 3. 133 3.5 Initiating a New Treatment 3. 134 CHAPTER 4: MISCELLANEOUS CONSIDERATIONS 4 135 4.1 Contacts by the Jaeb Center for Health Research and Sites 4 136 4.2 Subject Withdrawals 4 137 4.3 Management of Refractive Error 4 138 4.4 Risks 4 139 4.4.1 Risks of Examination Procedures 4 140 4.5 Reporting of Adverse Events 4 141 4.5.1 Risk Assessment 4 142 4.6 Discontinuation of Study 4 143 4.7 Travel Reimbursement 4 144 4.8 Study Costs 4 145 4.9 General Considerations 4 146 CHAPTER 5: SAMPLE SIZE ESTIMATION AND STATISTICAL ANALYSIS 5 147 5.1 Assessment of Investigator Interest / Recruitment Potential 5 148 | | 3.3.1 Follow-up Visit Testing Procedures for CI | 3-1 |
| 132 3.4 Non-study Visits 3. 133 3.5 Initiating a New Treatment 3. 134 CHAPTER 4: MISCELLANEOUS CONSIDERATIONS 4. 135 4.1 Contacts by the Jaeb Center for Health Research and Sites 4. 136 4.2 Subject Withdrawals 4. 137 4.3 Management of Refractive Error 4. 138 4.4 Risks 4. 139 4.4.1 Risks of Examination Procedures 4. 140 4.5 Reporting of Adverse Events 4. 141 4.5.1 Risk Assessment 4. 142 4.6 Discontinuation of Study 4. 143 4.7 Travel Reimbursement 4. 144 4.8 Study Costs 4. 145 4.9 General Considerations 4. 146 CHAPTER 5: SAMPLE SIZE ESTIMATION AND STATISTICAL ANALYSIS 5. 147 5.1 Assessment of Investigator Interest / Recruitment Potential 5. 148 5.2 Sample Size 5. 149 5.3 | | | |
| 133 3.5 Initiating a New Treatment 3. 134 CHAPTER 4: MISCELLANEOUS CONSIDERATIONS 4. 135 4.1 Contacts by the Jaeb Center for Health Research and Sites 4. 136 4.2 Subject Withdrawals 4. 137 4.3 Management of Refractive Error 4. 138 4.4 Risks 4. 139 4.4.1 Risks of Examination Procedures 4. 140 4.5 Reporting of Adverse Events 4. 141 4.5.1 Risk Assessment 4. 142 4.6 Discontinuation of Study 4. 143 4.7 Travel Reimbursement 4. 144 4.8 Study Costs 4. 145 4.9 General Considerations 4. 146 CHAPTER 5: SAMPLE SIZE ESTIMATION AND STATISTICAL ANALYSIS 5. 147 5.1 Assessment of Investigator Interest / Recruitment Potential 5. 148 5.2 Sample Size 5. 149 5.3 Primary Analysis – Symptom Success at One Year 5. 15 | 131 | 3.3.3 Follow-up Visit Testing Procedures for HT | 3-2 |
| 134 CHAPTER 4: MISCELLANEOUS CONSIDERATIONS | | 3.4 Non-study Visits | 3-2 |
| 135 4.1 Contacts by the Jaeb Center for Health Research and Sites 4 136 4.2 Subject Withdrawals 4 137 4.3 Management of Refractive Error 4 138 4.4 Risks 4 139 4.4.1 Risks of Examination Procedures 4 140 4.5 Reporting of Adverse Events 4 141 4.5.1 Risk Assessment 4 142 4.6 Discontinuation of Study 4 143 4.7 Travel Reimbursement 4 144 4.8 Study Costs 4 145 4.9 General Considerations 4 146 CHAPTER 5: SAMPLE SIZE ESTIMATION AND STATISTICAL ANALYSIS 5 147 5.1 Assessment of Investigator Interest / Recruitment Potential 5 148 5.2 Sample Size 5 149 5.3 Primary Analysis – Symptom Success at One Year 5 150 5.4 Secondary Analysis – Motor Success at One Year 5 | 133 | 3.5 Initiating a New Treatment | 3-2 |
| 136 4.2 Subject Withdrawals 4 137 4.3 Management of Refractive Error 4 138 4.4 Risks 4 139 4.4.1 Risks of Examination Procedures 4 140 4.5 Reporting of Adverse Events 4 141 4.5.1 Risk Assessment 4 142 4.6 Discontinuation of Study 4 143 4.7 Travel Reimbursement 4 144 4.8 Study Costs 4 145 4.9 General Considerations 4 146 CHAPTER 5: SAMPLE SIZE ESTIMATION AND STATISTICAL ANALYSIS 5 147 5.1 Assessment of Investigator Interest / Recruitment Potential 5 148 5.2 Sample Size 5 149 5.3 Primary Analysis – Symptom Success at One Year 5 150 5.4 Secondary Analysis – Motor Success at One Year 5 | | CHAPTER 4: MISCELLANEOUS CONSIDERATIONS | 4-1 |
| 137 4.3 Management of Refractive Error 4 138 4.4 Risks 4 139 4.4.1 Risks of Examination Procedures 4 140 4.5 Reporting of Adverse Events 4 141 4.5.1 Risk Assessment 4 142 4.6 Discontinuation of Study 4 143 4.7 Travel Reimbursement 4 144 4.8 Study Costs 4 145 4.9 General Considerations 4 146 CHAPTER 5: SAMPLE SIZE ESTIMATION AND STATISTICAL ANALYSIS 5 147 5.1 Assessment of Investigator Interest / Recruitment Potential 5 148 5.2 Sample Size 5 149 5.3 Primary Analysis – Symptom Success at One Year 5 150 5.4 Secondary Analysis – Motor Success at One Year 5 | 135 | | |
| 138 4.4 Risks 4 139 4.4.1 Risks of Examination Procedures 4 140 4.5 Reporting of Adverse Events 4 141 4.5.1 Risk Assessment 4 142 4.6 Discontinuation of Study 4 143 4.7 Travel Reimbursement 4 144 4.8 Study Costs 4 145 4.9 General Considerations 4 146 CHAPTER 5: SAMPLE SIZE ESTIMATION AND STATISTICAL ANALYSIS 5 147 5.1 Assessment of Investigator Interest / Recruitment Potential 5 148 5.2 Sample Size 5 149 5.3 Primary Analysis – Symptom Success at One Year 5 150 5.4 Secondary Analysis – Motor Success at One Year 5 | 136 | 4.2 Subject Withdrawals | 4-1 |
| 139 4.4.1 Risks of Examination Procedures 4 140 4.5 Reporting of Adverse Events 4 141 4.5.1 Risk Assessment 4 142 4.6 Discontinuation of Study 4 143 4.7 Travel Reimbursement 4 144 4.8 Study Costs 4 145 4.9 General Considerations 4 146 CHAPTER 5: SAMPLE SIZE ESTIMATION AND STATISTICAL ANALYSIS 5 147 5.1 Assessment of Investigator Interest / Recruitment Potential 5 148 5.2 Sample Size 5 149 5.3 Primary Analysis – Symptom Success at One Year 5 150 5.4 Secondary Analysis – Motor Success at One Year 5 | 137 | 4.3 Management of Refractive Error | 4-1 |
| 140 4.5 Reporting of Adverse Events 4 141 4.5.1 Risk Assessment 4 142 4.6 Discontinuation of Study 4 143 4.7 Travel Reimbursement 4 144 4.8 Study Costs 4 145 4.9 General Considerations 4 146 CHAPTER 5: SAMPLE SIZE ESTIMATION AND STATISTICAL ANALYSIS 5 147 5.1 Assessment of Investigator Interest / Recruitment Potential 5 148 5.2 Sample Size 5 149 5.3 Primary Analysis – Symptom Success at One Year 5 150 5.4 Secondary Analysis – Motor Success at One Year 5 | 138 | 4.4 Risks | 4-1 |
| 141 4.5.1 Risk Assessment 4. 142 4.6 Discontinuation of Study 4. 143 4.7 Travel Reimbursement 4. 144 4.8 Study Costs 4. 145 4.9 General Considerations 4. 146 CHAPTER 5: SAMPLE SIZE ESTIMATION AND STATISTICAL ANALYSIS 5. 147 5.1 Assessment of Investigator Interest / Recruitment Potential 5. 148 5.2 Sample Size 5. 149 5.3 Primary Analysis – Symptom Success at One Year 5. 150 5.4 Secondary Analysis – Motor Success at One Year 5. | 139 | 4.4.1 Risks of Examination Procedures | 4-1 |
| 141 4.5.1 Risk Assessment 4 142 4.6 Discontinuation of Study 4 143 4.7 Travel Reimbursement 4 144 4.8 Study Costs 4 145 4.9 General Considerations 4 146 CHAPTER 5: SAMPLE SIZE ESTIMATION AND STATISTICAL ANALYSIS 5 147 5.1 Assessment of Investigator Interest / Recruitment Potential 5 148 5.2 Sample Size 5 149 5.3 Primary Analysis – Symptom Success at One Year 5 150 5.4 Secondary Analysis – Motor Success at One Year 5 | 140 | 4.5 Reporting of Adverse Events | 4-1 |
| 143 4.7 Travel Reimbursement 4. 144 4.8 Study Costs 4. 145 4.9 General Considerations 4. 146 CHAPTER 5: SAMPLE SIZE ESTIMATION AND STATISTICAL ANALYSIS 5. 147 5.1 Assessment of Investigator Interest / Recruitment Potential 5. 148 5.2 Sample Size 5. 149 5.3 Primary Analysis – Symptom Success at One Year 5. 150 5.4 Secondary Analysis – Motor Success at One Year 5. | 141 | 4.5.1 Risk Assessment | 4-1 |
| 143 4.7 Travel Reimbursement 4. 144 4.8 Study Costs 4. 145 4.9 General Considerations 4. 146 CHAPTER 5: SAMPLE SIZE ESTIMATION AND STATISTICAL ANALYSIS 5. 147 5.1 Assessment of Investigator Interest / Recruitment Potential 5. 148 5.2 Sample Size 5. 149 5.3 Primary Analysis – Symptom Success at One Year 5. 150 5.4 Secondary Analysis – Motor Success at One Year 5. | 142 | 4.6 Discontinuation of Study | 4-1 |
| 144 4.8 Study Costs 4 145 4.9 General Considerations 4 146 CHAPTER 5: SAMPLE SIZE ESTIMATION AND STATISTICAL ANALYSIS 5 147 5.1 Assessment of Investigator Interest / Recruitment Potential 5 148 5.2 Sample Size 5 149 5.3 Primary Analysis – Symptom Success at One Year 5 150 5.4 Secondary Analysis – Motor Success at One Year 5 | 143 | | |
| 1454.9General Considerations4.146CHAPTER 5: SAMPLE SIZE ESTIMATION AND STATISTICAL ANALYSIS5.1475.1Assessment of Investigator Interest / Recruitment Potential5.1485.2Sample Size5.1495.3Primary Analysis – Symptom Success at One Year5.1505.4Secondary Analysis – Motor Success at One Year5. | | | |
| 146CHAPTER 5: SAMPLE SIZE ESTIMATION AND STATISTICAL ANALYSIS51475.1Assessment of Investigator Interest / Recruitment Potential51485.2Sample Size51495.3Primary Analysis – Symptom Success at One Year51505.4Secondary Analysis – Motor Success at One Year5 | 145 | · | |
| 1475.1Assessment of Investigator Interest / Recruitment Potential5.11485.2Sample Size5.11495.3Primary Analysis – Symptom Success at One Year5.11505.4Secondary Analysis – Motor Success at One Year5.1 | | | |
| 1485.2Sample Size5-1495.3Primary Analysis – Symptom Success at One Year5-1505.4Secondary Analysis – Motor Success at One Year5- | 147 | | |
| 149 5.3 Primary Analysis – Symptom Success at One Year | | | |
| 5.4 Secondary Analysis – Motor Success at One Year | | | |
| 151 5.5 Additional Analyses | 151 | | |
| 152 5.5.1 Secondary Outcomes at One Year | | | |
| 153 5.5.2 Outcomes at 10 Weeks | | · | |
| 154 CHAPTER 6: REFERENCES | | | |
| 155<br>155 | | | |

#### **CHAPTER 1: BACKGROUND AND SUMMARY**

This study is being conducted by the Pediatric Eye Disease Investigator Group (PEDIG) and is funded through a cooperative agreement from the National Eye Institute.

# 1.1 Background

# Epidemiology and clinical characteristics:

New onset adult strabismus has been estimated to affect 54.1/100,000 in a recent population-based study in the USA.<sup>1</sup> In this study, the most common types of new onset strabismus in adults, after paralytic strabismus, were convergence insufficiency (8.4/100,000), small angle hypertropia (7.5/100,000) and divergence insufficiency (6.0/100,000). For each of these types the incidence increased with increasing age.<sup>1</sup>

# **Convergence insufficiency:**

Convergence insufficiency (CI) is characterized by an exodeviation greater at near than at distance and a remote near point of convergence and/or decreased positive fusional vergence.<sup>2</sup> It is typically associated with symptoms such as diplopia, eyestrain, asthenopia, frontal headaches or problems reading.<sup>2-4</sup> Treatment consists of either exercises,<sup>3,4</sup>prisms,<sup>3,4</sup> surgery,<sup>4-6</sup> or botulinum toxin injection.<sup>7</sup>

There is a paucity of evidence for the effectiveness of treatment for CI in adults, with most previous reports studying effects in children. A recent Cochrane review<sup>2</sup> identified two previous randomized clinical trials in adults. Teitelbaum et al<sup>8</sup> randomly assigned 29 presbyopic patients with symptomatic CI to either progressive addition lenses with base-in prism or progressive addition lenses with no prism. The authors concluded that base-in prism glasses were effective in reducing the symptoms of CI, although interestingly, symptoms also significantly improved with progressive addition lenses with no prism.<sup>8</sup> Birnbaum et al<sup>9</sup> randomly assigned 60 male adult patients to receive office-based vision therapy/orthoptics with supplemental home therapy, home vision therapy alone, or no treatment. Office vision therapy with supplemental home therapy was reported to be most effective with a success rate of 62%. Despite the findings of these two randomized trials there remains much uncertainty as to which treatments are most effective for a given adult patient with CI and what are realistic success rates.

# **Divergence insufficiency:**

Divergence insufficiency (DI) esotropia is a comitant esodeviation worse at distance fixation than at near, typically associated with symptoms of diplopia at distance.<sup>10</sup> Treatment most often consists of either prism correction<sup>10-13</sup> or strabismus surgery.<sup>14, 15</sup> The established surgical procedure for DI esotropia is lateral rectus resection.<sup>16-18</sup> Nevertheless, in recent years bilateral medial rectus recession has been advocated.<sup>14, 15, 19</sup> There are few studies comparing treatments for DI esotropia, and little data on treatment outcomes, especially over the long-term. One recent study<sup>19</sup> claimed medial rectus recession was equivalent to lateral rectus resection but it was retrospective, not randomized, and had small sample size (n=24) and therefore of insufficient power to make such a determination.

#### Hypertropia:

- New onset small angle hypertropia (HT) in adults presents as a comitant hyperdeviation,
- 203 typically less than 10 prism diopters, in the absence of oblique muscle dysfunction. The patient

typically experiences symptoms of vertical diplopia. There are a range of possible causes for such vertical misalignment including skew deviation, sagging eye syndrome,<sup>20</sup> myotoxicity following cataract surgery,<sup>21,22</sup> presumed micro-vascular event, or even central peripheral rivalry (dragged fovea-diplopia syndrome).<sup>23-25</sup> Treatment most often consists of prism correction of diplopia or strabismus surgery, although partial occlusion may be used in cases of central peripheral rivalry. Regarding surgical approaches for small angle HT, some surgeons perform superior rectus recession, while others have advocated mini-tenotomy (snip) procedures.<sup>26</sup> There are, however, limited data on the effectiveness of these treatments for small angle HT and few studies, if any, comparing treatment outcomes.

### Prospective Observational Studies:

A prospective observational study monitors different forms of treatment applied to patients with a certain condition. Individuals are enrolled in a prospective observational study on the basis of either disease or exposure status. The care provider, not a protocol, decides how a patient gets treated. Through direct data collection from care providers, the results of the ongoing disease process and medical care can then be observed.

Prospective observational studies have the advantage of applying inclusion/exclusion criteria and not dictating management. The large patient sample often enables better estimation of outcome rates. Also, since data are collected within standard clinical practice, the results have high external validity. Weaknesses of observational studies include difficulty in identifying and controlling all sources of bias, and challenges with respect to data analyses. There may also be variability in time intervals between visits and treatments, and the potential for confounding makes treatment group comparisons difficult to interpret. Despite these weaknesses, future randomized controlled trials may be developed based on preliminary estimates of treatment effects that an observational study provides for the studied conditions.

#### 1.2 Rationale for the study

#### Purpose of an adult CI-DI-HT strabismus prospective observational study:

A prospective adult strabismus observational study will provide data on the numbers, types and clinical characteristics of adult patients with CI, DI or HT who are seen by PEDIG investigators and are receiving certain types of treatments, and on the outcomes of those treatments over one year. These data will be used to generate hypotheses for possible future PEDIG studies, including randomized trials. Data collected will include angle of deviation, diplopia severity, treatment type, and treatment outcome.

# Public health importance:

There are limited prospective, standardized data available on adults with convergence insufficiency, divergence insufficiency or small angle hypertropia, the commonest causes of non-paralytic adult strabismus. This study will inform regarding the numbers and types of adults with these conditions seen by PEDIG investigators, enabling the generation of hypotheses for potential PEDIG studies and estimation of their recruitment feasibility.

#### 1.3 Considerations

It is recognized that estimates of treatment success may be biased by patient selection, but for some conditions / treatments, these data will be the best available for planning future PEDIG studies.

1-2

# 252 1.4 Study Objectives

- 253 To describe clinical characteristics, treatments, and one-year outcomes of adults with
- 254 convergence insufficiency, divergence insufficiency, or small angle hypertropia. Treatment
- comparisons within the studied conditions will also be done to help develop future studies.

256257

- 1.5 Synopsis of Study Design
- 258 1.5.1 Synopsis of Study Design for CI
- 259 Major Eligibility Criteria (see section 2.2.1 for full details)
- Adults ≥18 years of age (adult onset of CI not required)
- No strabismus surgery in the past 10 years
- CI Symptom Survey score ≥21 points
- Near exodeviation of  $\geq 4\Delta$  and at least  $4\Delta$  larger than at distance by PACT
- Distance exodeviation ≤15Δ by PACT
- Vertical deviation  $\leq 2\Delta$  at distance and near by PACT
- No constant exotropia at distance or near
- Reduced positive fusional vergence (PFV) at near (<20Δ or fails Sheard's criterion that the PFV measures less than twice the magnitude of the near phoria)
- Near point of convergence (NPC) of ≥6 cm break
- No paralytic strabismus, paretic strabismus, restrictive strabismus, monocular diplopia,
- thyroid eye disease, myasthenia gravis, chronic progressive external ophthalmoplegia, or eye movement abnormalities associated with known neurological disease. Patients with
- 273 Parkinson's disease can be enrolled if non-paretic deviation.
- Visual acuity 20/50 or better in both eyes by ETDRS or Snellen
- Ability to fuse with prism in space (see section 2.4.1)
- Investigator is initiating treatment with prism, orthoptic exercises, botulinum toxin injection or surgery
- If initiating treatment with botulinum toxin or surgery, planned injection or surgery to be within 60 days of enrollment.
- Treatment to be initiated has not been used within the past one year

281

- 282 Treatment
- 283 Treatment is per the investigator's usual clinical practice.

284

- Data will be collected for the following treatment modalities:
- Bilateral medial rectus muscle resection surgery
- Single medial rectus muscle resection surgery
- Recess lateral rectus muscle resection medial rectus muscle surgery
- Bilateral lateral rectus muscle recession surgery
- Single lateral rectus muscle recession surgery
- Botulinum toxin injection
- 292 Prisms
- Orthoptic exercises, including computer-based therapy

294

- 295 Sample Size
- 296 50 subjects per non-surgical treatment modality (prism, orthoptic exercises) and up to 100
- subjects undergoing surgery (maximum 50 per surgical modality) will be enrolled, for a total of

up to 200 subjects with CI. Recruitment will continue for 1 year, at which time the determination will be made whether the recruitment period should be extended to allow for additional subjects to be enrolled in treatment modality groups that have not reached their maximum.

300 301 302

303

304

298

299

#### Visit Schedule

- Baseline Visit
- 10 week  $\pm$  3 weeks following intervention
- 12-months  $\pm$  2 months following intervention

305 306 307

308

309

Visits will be timed from the date of surgery or botulinum toxin injection (if applicable); or if prescribed prism or orthoptic exercises, visits will be timed from the day of enrollment. Subjects can remain in the study up to an additional year and have up to two additional follow up visits if their treatment modality is changed during the study.

310311

#### 312 Outcome

- The primary outcome will be symptom success at the 10-week and 12-month visit, defined as
- 314 improvement of CI Symptom Survey (CISS) score of at least 9 points and an outcome score of
- 315 <21 points. For surgical treatment, a secondary, motor outcome will evaluate how often subjects
- 316 have become orthotropic at distance and near after treatment.

317

### 1.5.2 Study Flow Chart: CI

319320

318

321

322323

324

#### **Baseline Exam**

#### Confirm Eligibility as Defined in Section 2.2.1

#### **Testing Procedures**

- CI Symptom Survey (CISS)
- Diplopia Questionnaire
- Adult Strabismus 20 (AS-20) Questionnaire
- Distance visual acuity (ETDRS or Snellen)
- Ocular Alignment (cover/uncover, SPCT, PACT)
- Fusion with prism in space
- Positive fusional vergence
- Near point of convergence

#### <u>Interim Outcome Exam: 10 weeks ± 3 weeks</u> <u>(timed from initiation of treatment)</u>

- CI Symptom Survey (CISS)
- Diplopia Questionnaire
- Adult Strabismus 20 (AS-20) Questionnaire
- Distance visual acuity (ETDRS or Snellen: Same as at baseline)
- Ocular Alignment (cover/uncover, SPCT, PACT)
- Positive fusional vergence
- Near point of convergence

#### <u>Outcome Exam: 12-Month ± 2 months exam</u> (timed from initiation of treatment)

- CI Symptom Survey (CISS)
- Diplopia Questionnaire
- Adult Strabismus 20 (AS-20) Questionnaire
- Distance visual acuity (ETDRS or Snellen: Same as at baseline)
- Ocular Alignment (cover/uncover, SPCT, PACT)
- Positive fusional vergence
- Near point of convergence

### 325 1.5.3 Synopsis of Study Design for DI

- 326 Major Eligibility Criteria (see section 2.2.2 for full details)
- Adults ≥18 years of age
- Adult-onset DI (at ≥18 years of age)
- No prior strabismus surgery
- Symptoms of diplopia at distance with a frequency of sometimes or worse in primary position
- Distance esodeviation of 2Δ to 30Δ and distance deviation is at least 1.25 times (25% larger than) near deviation by PACT (i.e., maximum near deviation is at least 20% smaller than distance deviation). The distance deviation must exceed the near deviation by at least the amounts provided in the table below.

336 337

**PACT Values for DI Eligibility** 

| Distance<br>Deviation | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 12 | 14 | 16 | 18 | 20 | 25 | 30 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| *Max Near<br>Deviation | 1 | 2 | 3 | 4 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 12 | 14 | 16 | 20 | 20 |

Calculation: Distance ≥ Near x 1.25 or Near ≤ Distance x 0.8

- No more than  $5\Delta$  difference between right and left gaze by PACT
- No more than 10Δ difference between primary position and either upgaze or downgaze by
   PACT
- Any coexisting vertical deviation must be less than the distance esodeviation and ≤10∆ by
   PACT
- No paralytic strabismus, paretic strabismus, restrictive strabismus, monocular diplopia,
   thyroid eye disease, myasthenia gravis, chronic progressive external ophthalmoplegia, or eye
   movement abnormalities associated with known neurological disease. Patients with
   Parkinson's disease can be enrolled if non-paretic deviation
- Visual acuity 20/50 or better in both eyes by ETDRS or Snellen
- Ability to fuse with prism in space (see section 2.4.2)
- Investigator is initiating treatment with prism, orthoptic exercises, botulinum toxin injection, or surgery
- If initiating treatment with botulinum toxin or surgery, planned injection or surgery to be within 60 days of enrollment.
- Treatment to be initiated has not been used within the past one year

357

#### 358 Treatment

359 Treatment is per the investigator's usual clinical practice.

- Data will be collected for the following treatment modalities:
- Bilateral lateral rectus muscle resection surgery
- Single lateral rectus muscle resection surgery
- Recess medial rectus muscle resection lateral rectus muscle surgery
- Bilateral medial rectus muscle recession surgery
- Single medial rectus muscle recession surgery
- Botulinum toxin injection

<sup>\*</sup>Near deviation is the nearest study-permitted prism based on Strabismus Procedures Manual.

- 368 Prisms
  - Orthoptic exercises, including computer-based therapy

369370

- 371 <u>Sample Size</u>
- 50 subjects per non-surgical treatment modality (prism, orthoptic exercises) and up to 150 subjects undergoing surgery (maximum 50 per surgical modality) will be enrolled, for a total of up to 250 subjects with DI. Recruitment will continue for 1 year, at which time the determination will be made whether the recruitment period should be extended to allow for additional subjects to be enrolled in treatment modality groups that have not reached their maximum.

378

- 379 <u>Visit Schedule</u>
- 380 Baseline Visit
  - 10 week  $\pm$  3 weeks following intervention
- 12-months  $\pm$  2 months following intervention

383 384

385

386

381

Visits will be timed from the date of surgery or botulinum toxin (if applicable); or if prescribed prism or orthoptic exercises, visits will be timed from the day of enrollment. Subjects can remain in the study up to an additional year and have up to two additional follow up visits if their treatment modality is changed during the study.

387 388 389

- Outcomes
- The primary outcome will be symptom success at the 10-week and 12-month visit, defined as diplopia "rarely" or "never" in primary position at distance on the diplopia questionnaire. For surgical treatment, a secondary, motor outcome will evaluate how often subjects have become orthotropic at distance and near after treatment.

# 1.5.4 Study Flow Chart: DI

396397

395

#### **Baseline Exam**

#### **Confirm Eligibility as Defined in Section 2.2.2**

#### **Testing Procedures**

- Diplopia Questionnaire
- Adult Strabismus 20 (AS-20) Questionnaire
- Distance visual acuity (ETDRS or Snellen)
- Ocular Alignment (cover/uncover, SPCT, PACT)
- Fusion with prism in space
- Negative fusional vergence

# <u>Interim Outcome Exam: 10 weeks ± 3 weeks</u> (timed from initiation of treatment)

- Diplopia Questionnaire
- Adult Strabismus 20 (AS-20) Questionnaire
- Distance visual acuity (ETDRS or Snellen: Same as at baseline)
- Ocular Alignment (cover/uncover, SPCT, PACT)
- Negative fusional vergence

# Outcome Exam: 12-Month ± 2 months exam (timed from initiation of treatment)

- Diplopia Questionnaire
- Adult Strabismus 20 (AS-20) Questionnaire
- Distance visual acuity (ETDRS or Snellen: Same as at baseline)
- Ocular Alignment (cover/uncover, SPCT, PACT)
- Negative fusional vergence

### 1.5.5 Synopsis of Study Design for HT

- 399 <u>Major Eligibility Criteria (see section 2.2.3 for full details)</u>
- Adults ≥18 years of age
- 401 Adult-onset HT (at  $\ge$ 18 years of age)
- No prior strabismus surgery
- Symptoms of diplopia at distance or near with a frequency of sometimes or worse in primary position at distance or reading position
- Vertical deviation  $\ge 1\Delta$  to  $\le 10\Delta$  at distance and near by prism and alternate cover test (PACT)
- No more than  $4\Delta$  difference from the primary in any gaze position by PACT
- Any coexisting esodeviation must be less than the vertical deviation by PACT
- 408 Any coexisting exodeviation ≤10 $\Delta$  by PACT
- No convergence insufficiency as defined in section 2.2.1
- No paralytic strabismus, paretic strabismus, restrictive strabismus, monocular diplopia, thyroid eye disease, myasthenia gravis, chronic progressive external ophthalmoplegia, or eye movement abnormalities associated with known neurological disease. Patients with
- Parkinson's disease can be enrolled if non-paretic deviation
- Visual acuity 20/50 or better in both eyes by ETDRS or Snellen
- Ability to fuse with prism in space (see section 2.4.3)
- Investigator is initiating treatment with prism, orthoptic exercises, botulinum toxin injection or surgery
- If initiating treatment with botulinum toxin or surgery, planned injection or surgery to be within 60 days of enrollment.
- Treatment to be initiated has not been used within the past one year

422 Treatment

Treatment is per the investigator's usual clinical practice.

424

421

398

- Data will be collected for the following treatment modalities:
- Vertical rectus muscle recession surgery
- Vertical rectus muscle mini-tenotomy (snip) surgery
- Botulinum toxin injection
- 429 Prisms
- Orthoptic exercises, including computer-based therapy

431

432 Sample Size

- 433 50 subjects per non-surgical treatment modality (prism, orthoptic exercises) and up to 100
- subjects undergoing surgery (maximum 50 per surgical modality) will be enrolled, for a total of
- 435 up to 200 subjects with HT. Recruitment will continue for 1 year, at which time the
- determination will be made whether the recruitment period should be extended to allow for
- additional subjects to be enrolled in treatment modality groups that have not reached their
- 438 maximum.

439

- 440 Visit Schedule
- 441 Baseline Visit
- 10-week  $\pm$  3 weeks following intervention
- 12-months  $\pm$  2 months following intervention

Visits will be timed from the date of surgery or botulinum toxin injection (if applicable); or if prescribed prism or orthoptic exercises, visits will be timed from the day of enrollment. Subjects can remain in the study up to an additional year and have up to two additional follow up visits if their treatment modality is changed during the study.

# 449450 Outcomes

 The primary outcome will be symptom success at the 10-week and 12-month visit, defined as diplopia "rarely" or "never" both in primary position at distance and in reading position on the diplopia questionnaire. For surgical treatment, a secondary, motor outcome will evaluate how often subjects have become orthotropic at distance and near after treatment.

### 1.5.6 Study Flow Chart: HT

457458

459

460

461

462

463

#### **Baseline Exam**

#### Confirm Eligibility as Defined in Section 2.2.3

#### **Testing Procedures**

- Diplopia Questionnaire
- Adult Strabismus 20 (AS-20) Questionnaire
- Distance visual acuity (ETDRS or Snellen)
- Ocular Alignment (cover/uncover, SPCT, PACT)
- Fusion with prism in space
- Vertical fusional amplitudes
- Double Maddox Rod Testing

# <u>Interim Outcome Exam: 10 weeks ± 3 weeks</u> (timed from initiation of treatment)

- Diplopia Questionnaire
- Adult Strabismus 20 (AS-20) Questionnaire
- Distance visual acuity (ETDRS or Snellen: Same as at baseline)
- Ocular Alignment (cover/uncover, SPCT, PACT)
- Vertical fusional amplitudes
- Double Maddox Rod Testing

#### <u>Outcome Exam: 12-Month ± 2 months exam</u> (timed from initiation of treatment)

- Diplopia Questionnaire
- Adult Strabismus 20 (AS-20) Questionnaire
- Distance visual acuity (ETDRS or Snellen: Same as at baseline)
- Ocular Alignment (cover/uncover, SPCT, PACT)
- Vertical fusional amplitudes
- Double Maddox Rod Testing

#### **CHAPTER 2: SUBJECT ENROLLMENT**

464 465

466

#### 2.1 **Eligibility Assessment and Informed Consent**

467 A maximum of 650 subjects will be enrolled in the study. A maximum of 50 subjects per 468 treatment modality (prism, orthoptic exercises, surgery of a specific type) per condition (CI, DI, 469

HT) will be enrolled, with up to 100 CI subjects treated with surgery, up to 150 DI subjects

470 treated with surgery, and up to 100 HT subjects treated with surgery. Recruitment will continue 471

for 1 year, at which time the determination will be made whether the recruitment period should

472 be extended to allow for additional subjects to be enrolled in treatment modality groups that have

473 not reached their maximum.

474 475

476

477

478

479

A subject is considered for the study after undergoing a routine eye examination (by a study investigator as part of standard of care), or a referral, that identifies CI, DI, or HT that appears to meet the eligibility criteria. The study will be discussed with the subject. Subjects who express an interest in the study will be given a copy of the informed consent form to read. Written informed consent must be obtained from the subject prior to performing any study-specific procedures that are not part of the subject's routine care.

480 481 482

483

484

486

506

#### 2.2 **Eligibility and Exclusion Criteria**

#### 2.2.1 **Eligibility Criteria for CI**

485 The following criteria must be met for the subject to be enrolled into the study:

- Adults ≥18 years of age (adult onset of CI not required)
- 487 No strabismus surgery within the past 10 years
- 488 CI Symptom Survey score ≥21 points
- 489 • Near exodeviation of  $\geq 4\Delta$  and at least  $4\Delta$  larger than at distance by PACT
- 490 Distance exodeviation  $\leq 15\Delta$  by PACT
- 491 • Vertical deviation  $\leq 2\Delta$  at distance and near by PACT
- 492 • No constant exotropia at distance or near
- 493 • Reduced positive fusional vergence (PFV) at near ( $<20\Delta$  or fails Sheard's criterion that the 494 PFV measures less than twice the magnitude of the near phoria)
- 495 Near point of convergence (NPC) of  $\geq 6$  cm break
- 496 Visual acuity 20/50 or better in both eyes by ETDRS or Snellen
- No paralytic strabismus (e.g., 3<sup>rd</sup>, 4<sup>th</sup>, or 6<sup>th</sup> cranial nerve palsies, skew deviation, Duane 497 498 syndrome)
- 499 • No restrictive strabismus (e.g., blowout fracture, thyroid eye disease, post scleral buckle, 500 Brown syndrome)
- 501 No monocular diplopia
- 502 No paretic strabismus, thyroid eye disease, myasthenia gravis, chronic progressive external 503 ophthalmoplegia, or eye movement abnormalities associated with known neurological 504 disease. Patients with Parkinson's disease can be enrolled if non-paretic deviation.
- 505 No inferior or superior oblique overaction defined as 2+ or greater
  - Ability to fuse with prism in space (see section 2.4.1)
- 507 Ability to understand and complete a survey
- 508 Investigator is initiating treatment with prism, orthoptic exercises, botulinum toxin injection 509 or surgery

- 510 • If initiating treatment with botulinum toxin or surgery, planned injection or surgery to be 511 within 60 days of enrollment
- 512 Single treatment modality is planned (e.g., no combined prism and orthoptic exercises)
- 513 Treatment to be initiated has not been used within the past one year

# 514 515

# 2.2.2 Eligibility Criteria for DI

- 516 The following criteria must be met for the subject to be enrolled into the study:
- 517 Adults ≥18 years of age
- 518 Adult-onset DI (at  $\geq$ 18 years of age)
- 519 No prior strabismus surgery
- 520 Symptoms of diplopia at distance with a frequency of sometimes or worse in primary position (in current glasses if wearing glasses) 521
- 522 Distance esodeviation of  $2\Delta$  to  $30\Delta$  and distance deviation is at least 1.25 times (25% larger 523 than) near deviation by PACT (i.e., maximum near deviation is at least 20% smaller than 524 distance deviation). The distance deviation must exceed the near deviation by at least the 525 amounts provided in the table below.

# 526

# 527

# **PACT Values for DI Eligibility**

| Distance<br>Deviation | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 12 | 14 | 16 | 18 | 20 | 25 | 30 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| *Max Near<br>Deviation | 1 | 2 | 3 | 4 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 12 | 14 | 16 | 20 | 20 |

Calculation: Distance ≥ Near x 1.25 or Near ≤ Distance x 0.8

# 529 530

528

- 531 • No more than  $5\Delta$  difference between right and left gaze by PACT
- No more than  $10\Delta$  difference between the primary position at distance and either upgaze or 532 533 downgaze  $\leq 10\Delta$  by PACT
- 534 • Any coexisting vertical deviation must be less than distance esodeviation and  $\leq 10\Delta$  by PACT
- Visual acuity 20/50 or better in both eyes by ETDRS or Snellen 535
- No paralytic strabismus (e.g., 3<sup>rd</sup>, 4<sup>th</sup>, or 6<sup>th</sup> cranial nerve palsies, skew deviation, Duane 536 537 syndrome)
- 538 • No restrictive strabismus (e.g., blowout fracture, thyroid eye disease, post scleral buckle, 539 Brown syndrome)
- 540 No monocular diplopia
- No paretic strabismus, thyroid eye disease, myasthenia gravis, chronic progressive external 541 542 ophthalmoplegia, or eye movement abnormalities associated with known neurological 543 disease. Patients with Parkinson's disease can be enrolled if non-paretic deviation
- 544 No inferior or superior oblique overaction defined as 2+ or greater
- 545 Ability to fuse with prism in space (see section 2.4.2)
- 546 Ability to understand and complete a survey
- 547 • Investigator is initiating treatment with prism, orthoptic exercises, botulinum toxin injection 548 or surgery
- 549 • If initiating treatment with botulinum toxin or surgery, planned injection or surgery to be 550 within 60 days of enrollment
- 551 Single treatment modality planned (e.g., no combined prism and orthoptic exercises)
- 552 Treatment to be initiated has not been used within the past one year

<sup>\*</sup>Near deviation is the nearest study-permitted prism based on Strabismus Procedures Manual.

553554

# 2.2.3 Eligibility Criteria for HT

- The following criteria must be met for the subject to be enrolled into the study:
- Adults ≥18 years of age
- Adult-onset HT (at  $\geq$ 18 years of age)
- No prior strabismus surgery
- Symptoms of diplopia at distance or near with a frequency of sometimes or worse in primary or reading position (in current glasses if wearing glasses)
- Vertical deviation  $\ge 1\Delta$  to  $\le 10\Delta$  at distance and near by PACT
- No more than  $4\Delta$  difference from the primary in any gaze position by PACT
- Any coexisting esodeviation must be less than the vertical deviation
- Any coexisting exodeviation ≤10 $\Delta$  by PACT
- No convergence insufficiency as defined in section 2.2.1
- Visual acuity 20/50 or better in both eyes by ETDRS or Snellen
- No paralytic strabismus (e.g., 3<sup>rd</sup>, 4<sup>th</sup>, or 6<sup>th</sup> cranial nerve palsies, skew deviation, Duane syndrome)
- No restrictive strabismus (e.g., blowout fracture, thyroid eye disease, post scleral buckle,
   Brown syndrome)
- No monocular diplopia
- No paretic strabismus, thyroid eye disease, myasthenia gravis, chronic progressive external
   ophthalmoplegia, or eye movement abnormalities associated with known neurological
   disease. Patients with Parkinson's disease can be enrolled if non-paretic deviation.
- No inferior or superior oblique overaction defined as 2+ or greater
- Ability to fuse with prism in space (see section 2.4.3)
- Ability to understand and complete a survey
- Investigator is initiating treatment with prism, orthoptic exercises, botulinum toxin injection or surgery
- If initiating treatment with botulinum toxin or surgery, planned injection or surgery to be within 60 days of enrollment
- Single treatment modality planned (e.g., no combined prism and orthoptic exercises)
- Treatment to be initiated has not been used within the past one year

584 585

586

587

588

#### 2.3 Historical Information

Historical information collected at enrollment will include the following:

- Presence of co-existing neurological conditions (e.g., Parkinson's, Progressive supranuclear palsy, basal ganglia disease, stroke, or intracranial tumor) and any treatment
- Presence of epiretinal membrane, age-related macular degeneration (dry or neovascular), or macular pathology (if known)
- Heart disease
- 592 Diabetes
- Autoimmune disease (other than myasthenia gravis and thyroid eye disease)
- Previous treatment for strabismus (surgical and/or non-surgical)
- Other major medical problems (e.g., significant head trauma)

#### 2.4 Procedures at the Enrollment Visit

All examination procedures must be tested before initiating planned treatment and within 7 days of enrollment. All examination procedures at enrollment are performed in the subject's current correction, if required, and without cycloplegia. Any subjects wearing pre-study prism correction will be measured in trial frames without prism (unless otherwise noted below). If new correction is prescribed on the day of testing, or if the subject forgot to bring his/her spectacles, then testing should be done in trial frames. Full details for each procedure are listed in the *Procedures Manual*.

#### 2.4.1 Enrollment Procedures for CI

1. Convergence Insufficiency Symptom Survey (CISS)

2. <u>Diplopia Questionnaire (DQ)</u>

3. Adult Strabismus 20 (AS-20) Questionnaire

4. <u>Distance Visual Acuity</u>

  Monocular distance visual acuity testing will be performed in each eye using ETDRS or Snellen optotypes.

 • If wearing ground-in prism correction, testing will be done wearing current correction with prism; if wearing Fresnel prism, testing will be done in trial frames without prism correction.

The following must be tested by an examiner who is a pediatric ophthalmologist, pediatric optometrist, or certified orthoptist.

5. Ocular Alignment Testing

 • Ocular alignment will be assessed by the cover/uncover test and by simultaneous prism and cover test (SPCT) in primary gaze position at distance (6 meters) and at near (1/3 meter).

 • Prism and alternate cover test (PACT) will be tested at distance (6 meters) and near (1/3 meter) in primary position.

6. <u>Fusion with Prism in Space</u>

 Ability to fuse with prism in space will be determined by asking the subject to view a 20/50 single optotype at 6 meters while neutralizing the deviation with free prisms. Subjects should be asked if they can make the image single. Subjects who are unable to make the image single are ineligible.

# 7. <u>Positive Fusional Vergence (PFV)</u>

 ■ PFV will be measured with a horizontal prism bar and a hand-held fixation target (20/50 single optotype) at 40 cm. Blur, break, and recovery points will be recorded. If no blur point is detected, the PFV score will be the break point measurement.

# 8. Near Point of Convergence (NPC)

• Break and recovery values will be measured.

| 212 | Enrollment | Procedures | for D |
|-------|------------|------------|-------|
| Z.4.Z | Enrollment | Procedures | TOP D |

# 1. <u>Diplopia Questionnaire</u>

# 2. Adult Strabismus 20 (AS-20) Questionnaire

### 3. Distance Visual Acuity

• Monocular distance visual acuity testing will be performed in each eye using ETDRS or Snellen optotypes.

 • If wearing ground-in prism correction, testing will be done wearing current correction with prism; if wearing Fresnel prism, testing will be done in trial frames without prism correction.

# The following must be tested by an examiner who is a pediatric ophthalmologist, pediatric optometrist, or certified orthoptist.

# 4. Ocular Alignment Testing

 • Ocular alignment will be assessed by the cover/uncover test and by simultaneous prism and cover test (SPCT) in primary gaze position at distance (6 meters) and at near (1/3 meter).

• Prism and alternate cover test (PACT) will be tested at distance (6 meters) and near (1/3 meter) in primary position.

# 5. Fusion with Prism in Space

 Ability to fuse with prism will be determined by asking the subject to view a 20/50 single optotype at 6 meters, and using prism(s), determine if any combination allows the subject to have single vision. Subjects who are unable to make the image single are ineligible.

# 6. Negative Fusional Vergence (NFV)

 NFV will be measured with a horizontal prism bar while the subject is viewing an accommodative target (20/50 single optotype) at 6 meters. Blur, break, and recovery points will be recorded. If no blur point is measured, the NFV score will be the break point measurement.

#### 2.4.3 Enrollment Procedures for HT

# 1. <u>Diplopia Questionnaire</u>

#### 2. Adult Strabismus 20 (AS-20) Questionnaire

#### 3. Distance Visual Acuity

 Monocular distance visual acuity testing will be performed in each eye using ETDRS or Snellen optotypes.

 • If wearing ground-in prism correction, testing will be done wearing current correction with prism; if wearing Fresnel prism, testing will be done in trial frames without prism correction.

The following must be tested by an examiner who is a pediatric ophthalmologist, pediatric optometrist, or certified orthoptist.

# 4. Ocular Alignment Testing

- Ocular alignment will be assessed by the cover/uncover test and by simultaneous prism and cover test (SPCT) in primary gaze position at distance (6 meters) and at near (1/3 meter).
- Prism and alternate cover test (PACT) will be tested at distance (6 meters) and near (1/3 meter) in primary position.

### 5. Fusion with Prism in Space

Ability to fuse with prism will be determined by asking the subject to view a 20/50 single optotype at 6 meters, and using prism(s), determine if any combination allows the subject to have single vision. Subjects who are unable to make the image single are ineligible.

# 6. <u>Vertical Fusional Amplitudes</u>

- Vertical fusional amplitudes will be measured with a vertical prism bar while the subject is viewing an accommodative target (20/50 single optotype) at 6 meters. Break and recovery points will be recorded. Measurements will be taken in both vertical directions to measure the range of vertical fusion.
- Vertical deviation should be corrected at least with sufficient prism to give the subject single vision either in current correction (if pre-study prism) or with prism correction in trial frames.

# 7. Double Maddox Rod Testing

• Ocular cyclotorsion will be assessed by double Maddox rod in primary gaze position at near (1/3 meters).

#### **CHAPTER 3: TREATMENT AND FOLLOW-UP**

723 724 725

#### 3.1 Treatment

- Treatment is at investigator discretion and may be changed or discontinued at any time during the study. The type of treatment and other treatment details (e.g., magnitude of prism, amount of orthoptic exercises) will be recorded at the time of enrollment when the treatment is prescribed.
- 729 For surgical subjects, the type and amount of surgery will be recorded. If an adjustable
- technique is used, the final location of the muscle and alignment after adjustment will be
- recorded. For those treated with botulinum toxin injection, the muscle(s) injected and dose will
- be recorded. The timing of surgical intervention after enrollment is at investigator discretion;
- however, the enrollment assessments must be redone if surgery is not done within 60 days.

734735

736

Changing treatment within a modality (e.g., frequency, strength, intensity) has no impact on the subject's visit schedule. Switching to a different treatment or adding a second treatment to the initial treatment has implications for the subject's visit schedule (see section 3.5).

737 738 739

# 3.2 Visit Schedule

Subjects enrolled will have visits at the following times:

- 10 weeks  $\pm$  3 weeks following intervention
- 12 months  $\pm$  2 months following intervention

743744

745

746

Visits will be timed from the date of surgery or botulinum toxin injection (if applicable); or if prescribed prism or orthoptic exercises, will be timed from the day of enrollment. If a new treatment is initiated, the visit schedule may restart or the subject's study participation may end, according to the details in *section 3.5*.

747 748 749

750

751

752

753

754

755

756

#### 3.3 Follow-up Visit Testing Procedures (10-week and 12-month visits)

At each visit, data on treatments received, any change in the amount/intensity of treatment, or any major change in eye condition since the last visit will be collected. In addition, the following will be performed / completed as done at the enrollment exam in the subject's current correction, if required, and without cycloplegia. Questionnaires and the symptom survey (if applicable) should be administered to the subject prior to other examination procedures. Any subjects wearing prism correction will be measured in trial frames without prism (unless otherwise noted below). If new correction is prescribed on the day of testing, or if the subject forgot to bring his/her spectacles, then testing should be done in trial frames.

757 758 759

761

762763

764

765

766

767

768

769

#### 3.3.1 Follow-up Visit Testing Procedures for CI

760 See section 2.4.1 for details.

- 1. CISS
- 2. Diplopia Questionnaire
- 3. AS-20 Questionnaire
- 4. Distance Visual Acuity
  - If wearing ground-in prism correction, testing will be done wearing current correction with prism; if wearing Fresnel prism, testing will be done in trial frames without prism correction.
- 5. Ocular Alignment Testing
- 6. Positive Fusional Vergence

7. Near Point of Convergence

# 3.3.2 Follow-up Visit Testing Procedures for DI

773 See section 2.4.2 for details.

- 1. Diplopia Questionnaire
- 2. AS-20 Questionnaire
- 3. Distance Visual Acuity
  - If wearing ground-in prism correction, testing will be done wearing current correction with prism; if wearing Fresnel prism, testing will be done in trial frames without prism correction.
- 4. Ocular Alignment Testing
- 781 5. Negative Fusional Vergence

# 3.3.3 Follow-up Visit Testing Procedures for HT

See *section 2.4.3* for details.

- 1. Diplopia Questionnaire
- 2. AS-20 Questionnaire
- 3. Distance Visual Acuity
  - If wearing ground-in prism correction, testing will be done wearing current correction with prism; if wearing Fresnel prism, testing will be done in trial frames without prism correction.
- 4. Ocular Alignment Testing
- 5. Vertical Fusional Amplitudes
  - Vertical deviation should be corrected at least with sufficient prism to give the subject single vision either in current correction (if pre-study prism) or with prism correction in trial frames.
- 6. Double Maddox Rod Testing

### 3.4 Non-study Visits

Additional non-study visits and treatment are at investigator discretion. Investigators must follow the procedures for initiating a new treatment during the study as outlined in *section 3.5*.

### 3.5 Initiating a New Treatment

If any new treatment is initiated during the study an early outcome exam as outlined in *section* 3.3 will be completed. Study participation will end if the new treatment is prism or exercises, unless initially enrolled in the surgery or botox injection group. If the new treatment is a new surgical modality or botox injection (not a re-operation or re-injection in the study), the examination will serve both as the outcome exam for the initial treatment and the baseline exam for the newly initiated surgery or botox injection, if the subject still meets eligibility criteria. The subject will then be followed for an additional 12-months in the study in the new treatment, as if they had been newly enrolled.

In the event that the study category for the newly initiated surgical modality is no longer recruiting subjects, the subject will complete an early outcome exam at the time the new surgery or botox injection is prescribed and study participation will end for this subject.

Subjects who have had surgery or botox injection as their initial treatment (or as a new treatment during the study) will continue to be followed until the 12-month outcome exam whether or not an additional treatment is initiated. The exception is if a re-operation or re-injection is planned prior to the 12-month outcome. In this case, an early outcome exam will be completed at the time surgery is prescribed. Study participation will end following the outcome examination.

Subjects who have completed the study and are returning for additional treatment following an unspecified period of time beyond the outcome exam may be enrolled a second time provided they meet eligibility criteria and the study category for the newly initiated treatment is still recruiting subjects. Subjects enrolling as a study subject a second time must repeat the consent process.

| 828<br>829 | | CHAPTER 4: MISCELLANEOUS CONSIDERATIONS |
|---|---|---|
| 830 | 4.1 | Contacts by the Jaeb Center for Health Research and Sites |
| 831<br>832<br>833<br>834<br>835<br>836<br>837 | with the before patient the Inc. | he be Center serves as the PEDIG Coordinating Center. The Jaeb Center will be provided the subject's contact information. The Jaeb Center will contact each subject one month any 12-month visit (including a second 12-month visit which could be required if the t changed treatments during the study). Permission for such contacts will be included in formed Consent Form. The principal purpose of the contacts will be to help coordinate uling of the 12-month outcome examination. |
| 838 | 4.2 | Subject Withdrawals |
| 839<br>840<br>841<br>842<br>843<br>844<br>845 | occurrindica<br>speak<br>eye ca | ets may withdraw from the study at any time. This is expected to be a very infrequent rence in view of the study design's similarity to routine clinical practice. If the subject tes they want to withdraw from the study, the investigator personally should attempt to with them to determine the reason. If their interest is in transferring their care to another are provider, every effort should be made to comply with this and at the same time try to the participant in the study under the new provider's care. |
| 846 | 4.3 | Management of Refractive Error |
| 847<br>848 | Manag | gement of refractive error is at the discretion of the investigator. |
| 849 | 4.4 | Risks |
| 850<br>851 | There | are no risks in this study that would not be part of usual care. |
| 852 | 4.4.1 | Risks of Examination Procedures |
| 853<br>854<br>855 | | rocedures in this study are part of daily eye care practice in the United States and pose no n risks. |
| 856 | 4.5 | Reporting of Adverse Events |
| 857<br>858<br>859 | | eatments are being prescribed that are not part of usual care. Investigators will abide by IRB reporting requirements. |
| 860 | 4.5.1 | Risk Assessment |
| 861<br>862<br>863 | | ne investigators' opinion that the protocol's level of risk is research not involving greater ninimal risk. |
| 864 | 4.6 | Discontinuation of Study |
| 865<br>866<br>867 | | nudy may be discontinued by the Steering Committee (with approval of the Data and Safety oring Committee) prior to the preplanned completion of enrollment and follow-up for all ets. |
| 868<br>869 | 4.7 | Travel Reimbursement |
| 870 | Subjec | cts will be compensated \$25 for each 10-week visit and \$50 for each 12-month visit (by |

SAS1 Protocol v2.0 4-11-16 4-1

money-card) up to a maximum of \$150. If there are extenuating circumstances, and the subject

is unable to complete study visits without additional funds for travel costs, additional funds may be provided.

874875

876

877

# 4.8 Study Costs

The study will pay for visits specific to the research study, but will not pay for usual care visits that would occur whether or not the subject was in the study. The cost of usual care visits will be the responsibility of the participant or his/her insurance company.

878879880

Any costs associated with treatment will not be paid for by the study and will be the responsibility of the participant or his/her insurance company.

881 882 883

#### 4.9 General Considerations

The study is being conducted in compliance with the policies described in the network policies document, with the ethical principles that have their origin in the Declaration of Helsinki, with the protocol described herein, and with the standards of Good Clinical Practice.

886 887 888

884

885

Data will be directly collected in electronic case report forms, which will be considered the source data.

889 890

- There is no restriction on the number of participants to be enrolled by a site. A risk-based
- 892 monitoring approach will be followed, consistent with the FDA "Guidance for Industry
- 893 Oversight of Clinical Investigations A Risk-Based Approach to Monitoring" (August 2013).

#### CHAPTER 5: SAMPLE SIZE ESTIMATION AND STATISTICAL ANALYSIS

#### 5.1 **Assessment of Investigator Interest / Recruitment Potential**

At the February 2014 PEDIG Study Group meeting, 18 (44%) of 41 ophthalmologist investigators and 26 (65%) of 40 optometrists investigators indicated they would be willing to participate in this study. In addition, 8 (20%) of 41 ophthalmologists and 8 (20%) of 40 optometrists rated this protocol in the top 5 of 18 protocol ideas reviewed with the group. The study ranked 13th among the 18 protocol ideas reviewed with the group for the 81 investigators overall.

Table 1 shows a summary of the results from a February 2015 email survey of PEDIG investigators. For each condition (CI, DI, and HT), investigators were asked whether they treated patients with the condition and how many they treated with various treatment modalities over the course of one year.

Table 1: Assessment of Recruitment Potential

| | Number of Patients Treated in One Year In PEDIG Network* | | |
|---|---|---|---|
| Condition | Prism | Orthoptic Exercises | Surgery |
| CI | 229 | 192 | 23** |
| DI | 119 | 20 | 85*** |
| HT | 194 | 10 | 39**** |

<sup>\*</sup> Cases treated with more than one type of treatment are counted for each type of treatment.

#### 5.2 Sample Size

The maximum total sample size of 650 is based on a convenience sample of a maximum of 50 subjects per treatment modality (prism, orthoptic exercises, surgery of a specific type) per condition (CI, DI, HT), with up to 100 subjects treated with surgery for CI and for HT, and up to 150 subjects treated with surgery for DI (Table 2).

Table 2: Maximum Sample Size for Each Condition/ Treatment Modality

| | | Maximum Sample Size | |
|-----------|-------|---------------------|---------|
| Condition | Prism | Orthoptic Exercises | Surgery |
| CI | 50 | 50 | 100* |
| DI | 50 | 50 | 150* |
| HT | 50 | 50 | 100* |

<sup>\*</sup>Within this limit for the total number of surgeries for a given condition, no more than 50 surgeries of a specific type (e.g. bilateral medial rectus recessions, bilateral lateral rectus resection, botulinum toxin injection, etc.) may be enrolled.

Based on the assessment of recruitment potential (section 5.1), about half of the modality/condition groups would be expected to be filled to 50 subjects within one year (see Table 1). The remaining modality/condition groups might have a smaller-than-desired sample size for analysis or might require recruitment for more than one year.

SAS1 Protocol v2.0 4-11-16 5-1

898 899 900

901

894

895 896

897

902 903 904

905 906 907

908

909

910

911 912

913 914

> 916 917

921

915

918 919 920

922 923

924 925 926

928 929

927

930

<sup>\*\*</sup> Bilateral medial rectus resection (N=11), other (N=12)

<sup>\*\*\*</sup> Bilateral medial rectus recession (N=51), bilateral lateral rectus resection (N=13), other (N=21)

<sup>\*\*\*\*</sup>Vertical rectus recession (N=37), other (N=2)

Table 3 shows the expected half-widths for the 95% confidence interval for the success proportion estimate for each modality/condition group.

Table 3: Expected ½-Width of 95% Confidence Interval as a Function of Sample Size and Success Proportion\*

| - | | | Sample S | ize | |
|---------------------------|-----|-----|----------|-----|-----|
| One-Year | | | | | |
| <b>Success Proportion</b> | 10 | 20 | 30 | 40 | 50 |
| 1% | 6% | 4% | 4% | 3% | 3% |
| 3% | 11% | 8% | 6% | 5% | 5% |
| 5% | 14% | 10% | 8% | 7% | 6% |
| 10% | 19% | 13% | 11% | 9% | 8% |
| 15% | 22% | 16% | 13% | 11% | 10% |
| 20% | 25% | 18% | 14% | 12% | 11% |
| 25% | 27% | 19% | 16% | 13% | 12% |
| 30% | 28% | 20% | 16% | 14% | 13% |
| 40% | 30% | 22% | 18% | 15% | 14% |
| 50% | 31% | 22% | 18% | 15% | 14% |

<sup>\*</sup>Note: The grey boxes indicate that validity of confidence interval widths is questionable because the normal approximation might not be valid given these low probability of success and/or small sample sizes.

After accounting for up to 5% loss to follow-up, a sample size of 50 patients per treatment modality (prism, orthoptic exercises, surgery of a specific type) per condition would contribute about 47 subjects to the point estimate for a dichotomous success/failure outcome at one year. With 47 subjects, the maximum width of the resulting confidence intervals on each point estimate would be  $\pm 14\%$ .

# 5.3 Primary Analysis – Symptom Success at One Year

For each of the modality/condition groups, the primary analysis will be an estimation of the proportion of patients of patients with treatment success based on improvement of symptoms at 10 weeks post intervention and at one year, with 95% confidence intervals.

Table 4 shows the criteria for symptom success for each condition, which will be used to assess all treatment modalities.

Table 4: One-Year Symptom Success Criteria for Each Condition

| Condition | One-Year Symptom Success Criteria |
|---|---|
| CI | improvement of CI Symptom Survey (CISS) score of at least 9 points AND a |
| | score of <21 points |
| DI | diplopia no more than rarely in the past week in the primary position (question |
| | #1.1 on the Diplopia questionnaire) |
| HT | diplopia no more than rarely in the past week both in the primary position and |
| | for reading (questions #1.1 and #1.2 on the Diplopia questionnaire) |

For patients who initiate a new treatment before completing one year of follow-up, the symptom success/failure status from the visit at which treatment was changed (i.e., the 10-week interim visit or an early outcome visit) will be brought forward as their one-year outcome.

Rubin's multiple imputation<sup>21</sup> will be used to impute outcome for patients who have not changed treatments but who are who are lost to follow-up or withdraw from the study prior to one-year exam.

# 5.4 Secondary Analysis – Motor Success at One Year

For each surgery type within a condition, a secondary objective will be to calculate the proportion of patients with motor success at one year and a 95% confidence interval. Motor success will be defined as orthotropia by cover/uncover at distance and near fixation in primary position at one year. Similar to the primary analysis of symptom success, for patients who change treatments before completing one year of follow-up, the motor success/failure status from the visit at which treatment was changed (i.e., the 10-week interim visit or an early outcome visit) will be brought forward as the one-year outcome. In addition, Rubin's multiple imputation<sup>21</sup> will be used to impute outcome for patients who have not changed treatments but who are who are lost to follow-up or withdraw from the study prior to one-year exam.

### 5.5 Additional Analyses

## 5.5.1 Secondary Outcomes at One Year

Secondary outcomes at one year will be evaluated within each modality/condition. Secondary outcomes to be assessed include motor alignment, near point of convergence (CI only), positive fusional vergence (CI only), negative fusional vergence (DI only), vertical fusional vergence (HT only), and the Adult Strabismus 20 (AS-20) questionnaire. In addition, mean CI Symptom Survey (CISS) score will be evaluated for CI, and the AS-20 and Diplopia Questionnaire will be evaluated as a continuous outcomes for all three conditions.

# 5.5.2 Outcomes at 10 Weeks

Outcomes at the 10-week interim visit will be evaluated similarly to the primary and secondary analyses defined for one-year time points (sections 5.3, 5.4 and 5.5.1).

#### **CHAPTER 6: REFERENCES**

989 990

- 991 1. Martinez-Thompson JM, Diehl NN, Holmes JM, Mohney BG. Incidence, types, and lifetime risk of adult-onset strabismus. *Ophthalmology* 2014;121:877-882.
- Scheiman M, Gwiazda J, Li T. Non-surgical interventions for convergence insufficiency.
   Cochrane Database of Systematic Reviews 2011;16:CD006768.
- 3. Lavrich JB. Convergence insufficiency and its current treatment. *Current Opinion in Ophthalmology* 2010;21:356-360.
- 4. Cooper J, Jamal N. Convergence insufficiency-a major review. *Optometry* 2012;83:137-158.
- 5. von Noorden GK. Resection of both medial rectus muscles in organic convergence insufficiency. *American Journal of Ophthalmology* 1976;81:223-226.
- 1000 6. Choi DG, Rosenbaum AL. Medial rectus resection(s) with adjustable suture for intermittent exotropia of the convergence insufficiency type. *Journal of AAPOS: American Association* 1002 for Pediatric Ophthalmology & Strabismus 2001;5:13-17.
- 7. Saunte JP, Holmes JM. Sustained improvement of reading symptoms following botulinum toxin A injection for convergence insufficiency. *Strabismus* 2014;22:95-99.
- 1005 8. Teitelbaum B, Pang Y, Krall J. Effectiveness of base in prism for presbyopes with convergence insufficiency. *Optometry and Vision Science* 2009;86:153-156.
- 1007
   9. Birnbaum MH, Soden R, Cohen AH. Efficacy of vision therapy for convergence
   1008 insufficiency in an adult male population. *Journal of the American Optometric Association* 1009 1999;70:225-232.
- 1010 10. Scheiman M, Gallaway M, Ciner E. Divergence insufficiency: characteristics, diagnosis, and treatment. *American Journal of Optometry & Physiological Optics* 1986;63:425-431.
- 1012 11. Tamhankar MA, Ying GS, Volpe NJ. Effectiveness of prisms in the management of diplopia
   1013 in patients due to diverse etiologies. *Journal of Pediatric Ophthalmology and Strabismus* 1014 2012;49:222-228.
- 1015 12. Prangen Ade H, Koch FL. Divergence Insufficiency: A Clinical Study. *Transactions of the American Ophthalmological Society* 1937;35:136-148.
- 1017 13. Godts D, Mathysen DG. Distance esotropia in the elderly. *British Journal of Ophthalmology* 2013;97:1415-1419.
- 1019 14. Thomas AH. Divergence insufficiency. *Journal of AAPOS: American Association for Pediatric Ophthalmology & Strabismus* 2000;4:359-361.
- 15. Bothun ED, Archer SM. Bilateral medial rectus muscle recession for divergence insufficiency pattern esotropia. *Journal of AAPOS: American Association for Pediatric Ophthalmology & Strabismus* 2005;9:3-6.
- 1024 16. Wiggins RE, Jr., Baumgartner S. Diagnosis and management of divergence weakness in adults. *Ophthalmology* 1999;106:1353-1356.
- 1026 17. Simpson GV. Primary divergence insufficiency. *Transactions of the American Ophthalmological Society* 1973;71:152-161; discussions 161-152.
- 18. Stager DR, Sr., Black T, Felius J. Unilateral lateral rectus resection for horizontal diplopia in adults with divergence insufficiency. *Graefes Archive for Clinical and Experimental Ophthalmology* 2013;251:1641-1644.
- 19. Chaudhuri Z, Demer JL. Medial rectus recession is as effective as lateral rectus resection in divergence paralysis esotropia. *Archives of Ophthalmology* 2012;130:1280-1284.
- 20. Chaudhuri Z, Demer JL. Sagging eye syndrome: connective tissue involution as a cause of horizontal and vertical strabismus in older patients. *JAMA Ophthalmology* 2013;131:619-625.
- 1036 21. Rainin EA, Carlson BM. Postoperative diplopia and ptosis. A clinical hypothesis based on the myotoxicity of local anesthetics. *Archives of Ophthalmology* 1985;103:1337-1339.

- 1038 22. Johnson DA. Persistent vertical binocular diplopia after cataract surgery. *American Journal of Ophthalmology* 2001;132:831-835.
- 1040 23. Burgess D, Roper-Hall G, Burde RM. Binocular diplopia associated with subretinal neovascular membranes. *Archives of Ophthalmology* 1980;98:311-317.
- 1042 24. Brazis PW, Lee AG, Bolling JP. Binocular vertical diplopia due to subretinal neovascular membrane. *Strabismus* 1998;6:127-131.
- 25. De Pool ME, Campbell JP, Broome SO, Guyton DL. The dragged-fovea diplopia syndrome: clinical characteristics, diagnosis, and treatment. *Ophthalmology* 2005;112:1455-1462.
- 1046 26. Wright KW. Mini-tenotomy procedure to correct diplopia associated with small-angle strabismus. *Transactions of the American Ophthalmological Society* 2009;107:97-102. 1048